CLINICAL TRIAL: NCT04189250
Title: Comparison of the Automatized and the Optimized Carbon Monoxid Rebreathing Protocol Determining Hemoglobinmass With Capillary and Venous Blood Sampling
Brief Title: Comparison of the Automatized and the Optimized Carbon Monoxid Rebreathing Protocol
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Swiss Federal Institute of Sport Magglingen (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: COMP_aCO_oCO
Record Dates: First submitted 2019-12-03; First posted 2019-12-06 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hemoglobins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimized carbonmonoxid rebreathing protocol (oCO) (Placebo Comparator): 2 min rebreathing period seated position capillary blood sampling
  Interventions: Device: Automatized carbonmonoxide rebreathing machine - OpCO Detalo instruments
- Automatized carbonmonoxide rebreathing protocol (aCO) (Active Comparator): 10 minutes rebreathing period supine position venous blood sampling
  Interventions: Device: Automatized carbonmonoxide rebreathing machine - OpCO Detalo instruments

INTERVENTIONS:
Device: Automatized carbonmonoxide rebreathing machine - OpCO Detalo instruments — The automatized protocol (aCO) will be conducted with automated system OpCO of Detalo instruments. The intended use of the OpCO Detalo instrument is to quantify hemoglobin mass in human. The principle behind the machine is the widely used CO rebreathing technique. The machine applies automatically the desired CO dose to the patient to determine hemoglobin mass. The Detalo Instruments OpCO is certified conform to the following CE norms: Electromagentic compabilitiy: DIN EN 60601-1-2 and electrical Safety test: LVD 2014/35/EU.

SUMMARY:
The aim of this study is the comparison of two measurement protocols determining hemoglobin mass with two different blood sampling strategies.Both protocols are based on the principle of the carbonmonoxid (CO) rebreathing method. During this measurement, CO is inhaled for a specific time period by the subject in a closed circuit and it is used as a marker to tag circulating hemoglobin.

DETAILED DESCRIPTION:
The optimized CO rebreathing protocol (oCO) will be compared against the automatized CO rebreathing protocol (aCO). Although theses two protocols using the same method, they show some relevant differences.

The oCO use a 2 minutes rebreathing period in a seated position and capillary blood is taken. The aCO use a 10 minutes rebreathing period in a supine position and venous blood samples are taken.

It is essential to know to what extent the aCO with capillary or venous blood sampling with different rebreathing time and position compared to oCO will influence the provided hemoglobin mass values. It is important to ensure the comparability of formely hemoglobinmass data measured using oCO with hemoglobinmass data measured using aCO for scientific research.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or higher
* healthy (self-reported)
* women and men

Exclusion Criteria:

* smoker
* implementation of high altitude training six weeks before and during the study
* sickness before and during the study
* blood donation 6 weeks before and during the study
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-04-20 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of two CO rebreathing protocols (aCO and oCO) | During data collection (3 months)
  The aim is to assess the confidence interval of aCO with a ten min rebreathing period in supine position compared to oCO with a two min seated rebreathing period. The mean difference in hemoglobin mass will be determined, using the aCO and oCO.
Comparison of capillary and venous bloodsampling | During data collection (3 months)
  The aim is to compare capillary and venous blood samples collected simultaneously during aCO. The goal is to determine, if the site of blood sampling alters the measured carboxy-hemoglobin and hence the calculated hemoglobin mass.
  The outcome will be the confidence interval of mean difference measured with capillary and venous blood sampling.

SECONDARY OUTCOMES:
Reliability of aCO and oCO | During data collection (3 months)
  The aim is the determination of the reliability of aCO and oCO by implementing double measurements for both protocols. The coefficient of variation (CV) of hemoglobin mass measured for aCO and oCO will be a further outcome of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Wehrlin, Dr. scient., MSc., Principal Investigator — Swiss Federal Institute of Sport Magglingen
Locations (1):
- Swiss Federal Instistiution of Sport, Magglingen, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidt W, Prommer N. The optimised CO-rebreathing method: a new tool to determine total haemoglobin mass routinely. Eur J Appl Physiol. 2005 Dec;95(5-6):486-95. doi: 10.1007/s00421-005-0050-3. Epub 2005 Oct 13. PMID 16222540
- [Background] Fagoni N, Breenfeldt Andersen A, Oberholzer L, Haider T, Meinild Lundby AK, Lundby C. Reliability and validity of non-invasive determined haemoglobin mass and blood volumes. Clin Physiol Funct Imaging. 2018 Mar;38(2):240-245. doi: 10.1111/cpf.12406. Epub 2017 Jan 30. PMID 28135764
- [Background] Siebenmann C, Keiser S, Robach P, Lundby C. CORP: The assessment of total hemoglobin mass by carbon monoxide rebreathing. J Appl Physiol (1985). 2017 Sep 1;123(3):645-654. doi: 10.1152/japplphysiol.00185.2017. Epub 2017 Jun 29. PMID 28663373
- [Background] Steiner T, Wehrlin JP. Comparability of haemoglobin mass measured with different carbon monoxide-based rebreathing procedures and calculations. Scand J Clin Lab Invest. 2011 Feb;71(1):19-29. doi: 10.3109/00365513.2010.534174. Epub 2010 Nov 23. PMID 21091271